CLINICAL TRIAL: NCT01002612
Title: Reassessment of the Nutritional Status in Thai Orphans Living With HIV in a Family Style Community: 6 Months After Nutrition Care Support by the Thai-Australian Collaboration HIV-Nutrition (TACHIN) Project
Brief Title: Reassessment of the Nutritional Status in Thai Orphans Living With HIV in a Family Style Community
Acronym: TACHIN003-1
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Mahidol University (Other); South Eastern Area Health Service (Other)
Responsible Party: Supabhorn Pengnonyang, Nurse Nutritionist, Thai Red Cross AIDS Research Centre
Other Study IDs: TACHIN003.1
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infection; HIV Infections
Keywords: Nutritional status; Thai HIV-infected children
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To reassess nutritional status of HIV-infected Thai children living in the family style community after receiving nutrition support program for 6 months.

DETAILED DESCRIPTION:
The first assessment indicated that improving dietary intake, either energy or micronutrient intakes, to meet the recommended for HIV-infected children (CLHIV) would be able to improve growth of these children. We implemented the nutrition support program through the two strategies aiming to increase dietary intake for all children to meet the current World Health Organization (WHO) recommendations which the recommended energy requirements are increased by10% for asymptomatic CLHIV and increased by 20 to 50% for children who require catch up growth or experiencing opportunistic infections. The nutrition support program composed two strategies. Firstly is providing nutrition education to caregivers and also children. Secondly, revision food menus by caregivers with assisting from the nutritionists of the project. After this program have been implemented for 6 months, reassessment is needed to evaluate the changes of nutritional status and health outcomes in this children aiming to further providing support and applying to other settings.

ELIGIBILITY:
Inclusion Criteria:

* Children age 4-15 years old
* Confirmed HIV-1 diagnosis
* Reside at the community
* The guardian must be able and willing to provide written informed consent. Oral consent in the presence of witness is acceptable in the case of illiteracy

Exclusion Criteria:

* non-HIV infected children
* Age 0-3 years

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thai HIV-infected children living in a family style community located in rural central region of Thailand
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Growth parameters (weight and height), blood lipid levels and dietary intakes | 6 months

SECONDARY OUTCOMES:
Morbidity, CD4, HIV-RNA and satisfaction of caregivers and children | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, Principal Investigator — The Thai Red Cross AIDS Research Centre
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathumwan, Bangkok, Thailand